CLINICAL TRIAL: NCT03006107
Title: Comparison of the Efficacy of Prophylactic Intraligamentary Injection of Piroxicam Versus Mepecaine for Management of Post-endodontic Pain in Posterior Teeth
Brief Title: Comparison of a Prophylactic Intraligamentary Injection of Piroxicam Versus Mepecaine of Post-endodontic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Gamal Ahmed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: piroxicam _ Mepecaine
Record Dates: First submitted 2016-12-15; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Pulpitis - Irreversible
Keywords: Irreversible pulpitis; Post endodontic pain; Symptomatic pulpitis pain; Single visit RCT pain; Root canal treatment flare up; Single dose piroxicam; Intraligamentary piroxicam; Intraligamentary mepecaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intraligamentary injection of piroxicam (Experimental): intraligamentary injection Piroxicam is another NSAID that which has the ability for the treatment of pain, fever and inflammation in the body , has a half-life of 50h in the plasma , oral piroxicam reaches a peak concentration in the plasma within 2 to 4 hours .
  The needle will be placed in the gingival sulcus at a 30- degree angle to the long axis of the tooth then apical pressure is applied until the needle wedged into the periodontal ligament between the tooth and the alveolar crest of the bone
  Interventions: Procedure: intraligamentary injection piroxicam
- Intraligamentary mepevacaine (Active Comparator): mepevacaine is an anesthetic (numbing medicine) that blocks the nerve impulses that send pain signals to brain . It is also used as an anesthetic for dental procedures.
  Interventions: Procedure: Intraligamentary mepevacaine

INTERVENTIONS:
Procedure: intraligamentary injection piroxicam — intraligamentary injection Piroxicam is another NSAID that which has the ability for the treatment of pain, fever and inflammation in the body , has a half-life of 50h in the plasma , oral piroxicam reaches a peak concentration in the plasma within 2 to 4 hours .
  The needle will be placed in the gingival sulcus at a 30- degree angle to the long axis of the tooth then apical pressure is applied until the needle wedged into the periodontal ligament between the tooth and the alveolar crest of the bone
  Arms: intraligamentary injection of piroxicam
Procedure: Intraligamentary mepevacaine — mepevacaine is an anesthetic (numbing medicine) that blocks the nerve impulses that send pain signals to brain . It is also used as an anesthetic for dental procedures.
  Arms: Intraligamentary mepevacaine

SUMMARY:
to evaluate the effect of a single intraligamentary injection of piroxicam on postoperative pain associated with endodontic procedures.

DETAILED DESCRIPTION:
The pain after endodontic treatment is commonly severe in the first 24 hours after treatment, then it will reduce gradually until commonly disappearing after 7-10 days in most cases. Since piroxicam has a half-life of 50 hours in the plasma, it will be effective in controlling the most intense pain which occurs after endodontic treatment It appears that optimal clinical benefits can be achieved by administering drugs such as local anesthetics and NSAIDs before the onset of postoperative pain. Administering these drugs before a surgical or an endodontic procedure may be of benefit for longer procedures or for minimizing peripheral sensitization, which is a result of the cascade of inflammatory mediators that are released by tissue injury and fuel the subsequent inflammatory process

ELIGIBILITY:
Inclusion Criteria:

* • Medically free patients

  * Patient's age between 25-50 years.
  * Molar or premolar teeth diagnosed clinically and radiographically with irreversible pulpitis and symptomatic apical periodontitis.
  * Positive patient's acceptance for participation in the study.
  * Sex include both male and female.
  * Patients who can understand Numerical Rating Scale (NRS)
  * Patients able to sign informed consent.

Exclusion Criteria:

* • Pregnancy or lactation in female patients

  * Medically compromised patients.
  * Patient with multiple teeth that required endodontic treatment to eliminate the possibility of pain referral.
  * Patient with fracture or mobile or mutilated teeth.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-11 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The degree of postoperative pain at 6, 12, 24 and 48 postoperative hours which will be measured by Numeric Rate Scale , where the patient will be asked to rate the progress of pain on the NRS and inform the investigator with the results. | up to 48 hours
  Primary outcome will be collected by the operator through Numerical Rating Scale (NRS)20 which is an 11-point scale consisting of numbers from 0 through 10; 0 reading represents "no pain" , 1- 3 readings represent "mild pain" , 4- 6 readings represent "moderate pain" , 7- 10 readings represent "severe pain" No or mild pain will be considered as success while moderate or severe pain will be regarded as failure.

CONTACTS AND LOCATIONS:
Overall Officials: Angie g Ghoneim, Professor, Study Chair — Department of endodontics - Faculty of Oral and Dental medicine - CU; marwa ga ahmed, student, Principal Investigator — Department of endodontics - Faculty of Oral and Dental medicine - CU

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Penniston SG, Hargreaves KM. Evaluation of periapical injection of Ketorolac for management of endodontic pain. J Endod. 1996 Feb;22(2):55-9. doi: 10.1016/S0099-2399(96)80272-X. PMID 8935018
- [Background] Pharmacological Strategies to Control Post-operative Endodontic Pain. Dental Research Journal (Vol. 4, No. 2, Autumn-Winter 2007
- [Background] 3. Building effective strategies for the management of endodontic pain. Endodontic Topics 2002, 3, 93-105
- [Background] Atbaei A, Mortazavi N. Prophylactic intraligamentary injection of piroxicam (feldene) for the management of post-endodontic pain in molar teeth with irreversible pulpitis. Aust Endod J. 2012 Apr;38(1):31-5. doi: 10.1111/j.1747-4477.2010.00274.x. Epub 2010 Oct 24. PMID 22432824
- [Background] Torabinejad M, Bakland LK. Prostaglandins: their possible role in the pathogenesis of pulpal and periapical diseases, part 2. J Endod. 1980 Oct;6(10):769-76. doi: 10.1016/S0099-2399(80)80107-5. No abstract available. PMID 7005368
- [Background] Cohen JS, Reader A, Fertel R, Beck M, Meyers WJ. A radioimmunoassay determination of the concentrations of prostaglandins E2 and F2alpha in painful and asymptomatic human dental pulps. J Endod. 1985 Aug;11(8):330-5. doi: 10.1016/s0099-2399(85)80039-x. No abstract available. PMID 3863874
- [Background] McNicholas S, Torabinejad M, Blankenship J, Bakland L. The concentration of prostaglandin E2 in human periradicular lesions. J Endod. 1991 Mar;17(3):97-100. doi: 10.1016/S0099-2399(06)81737-1. PMID 1940730
- [Background] Mehrvarzfar P, Abbott PV, Saghiri MA, Delvarani A, Asgar K, Lotfi M, Karamifar K, Kharazifard MJ, Khabazi H. Effects of three oral analgesics on postoperative pain following root canal preparation: a controlled clinical trial. Int Endod J. 2012 Jan;45(1):76-82. doi: 10.1111/j.1365-2591.2011.01950.x. Epub 2011 Sep 8. PMID 21902704
- [Background] Mehlisch DR. The efficacy of combination analgesic therapy in relieving dental pain. J Am Dent Assoc. 2002 Jul;133(7):861-71. doi: 10.14219/jada.archive.2002.0300. PMID 12148679
- [Background] Maccagno A, Di Giorgio EE, Caston OL, Sagasta CL. Double-blind controlled clinical trial of oral S-adenosylmethionine versus piroxicam in knee osteoarthritis. Am J Med. 1987 Nov 20;83(5A):72-7. doi: 10.1016/0002-9343(87)90855-2. PMID 3318443